CLINICAL TRIAL: NCT06503848
Title: Migraine Attack Treatment Response Molecular and Clinical BiOmarkers (The MAMBO Study) Phase I
Brief Title: Migraine Attack Treatment Response Molecular and Clinical BiOmarkers (MAMBO) Phase I
Acronym: MAMBO
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: EOM(AG)053/2022(6055)
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Migraine Disorders
Keywords: migraine; triptan
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- episodic migraine: Patients with episodic migraine will be asked to treat four spontaneous migraine attacks with sumatriptan 50 milligrams. They will register the headache characteristics and whether or not the treatment was effective.
  Interventions: Drug: Sumatriptan

INTERVENTIONS:
Drug: Sumatriptan — Register the response to treatment and headache characteristics.

SUMMARY:
The goal of this observational study is to identify differential traits in spontaneous migraine attacks that can help us predict the response to treatment with sumatriptan.

Participants will be asked to register the headache characteristics before and after taking sumatriptan and whether the treatment was effective or not during four migraine attacks.

DETAILED DESCRIPTION:
There is still an unmet need in acute migraine treatment, some patients don't respond properly to acute medication.

There are some interindividual differences in clinical characteristics of migraine attacks. These differences may determine the response to acute treatment. Describing the phenotypical differences between patients who are responders and patients non-responders will allow us to offer a personalized treatment.

The aim of the study is to determine which characteristics are associated with a response or a non-response to acute treatment with sumatriptan.

Participants will be asked to register the headache characteristics and accompanying symptoms during 4 spontaneous migraine attacks and its response to treatment with sumatriptan.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with or without aura diagnosis according to ICHD-3 criteria
* <8 migraine days per month
* Be able to read, write and understand instructions.
* Have internet access and mail address
* Signing of the informed consent

Exclusion Criteria:

* Active preventive treatment for migraine
* Active medication with an effect over the central nervous system
* Serious physical or psychiatric condition
* Cardiovascular or hepatic disease
* Pregnant or breastfeeding women
* Any triptan contraindication
* Severe migraine attacks without previous response to triptans or NSAIDs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Otherwise healthy episodic migraine patients.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Response to sumatriptan | 24 hours
  Relief of pain from moderate-severe to mild or absent at 2 hours and 24 hours in 3 out of 4 migraine attacks.
  The response will be evaluated via questionnaire.

SECONDARY OUTCOMES:
Migraine characteristics | 24 hours
  Patients will complete a questionnaire describing the characteristics of migraine attacks in the beginning of the attack, and at timepoints 2 and 24 hours after taking sumatriptan.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Torres-Ferrús, PhD, Principal Investigator — Hospital Universitari Vall d'Hebron, Headache & Neurological Pain Research Group
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided